CLINICAL TRIAL: NCT02759081
Title: A Randomized, Controlled Trial Comparing Cap-assisted Water Exchange and Water Exchange in Colonoscopy
Brief Title: Comparing Cap-assisted Water Exchange and Water Exchange in Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hsi hsieh, Chief of endoscopy suite, deparment of Gastroenterology, Dalin Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Hsieh-2016-01
Record Dates: First submitted 2016-04-05; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Colonoscopy; Intubation Time; Cap-assisted Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water exchange (Active Comparator): The air was turned off at the beginning of colonoscopy. Water was infused and suctioned at the same time during insertion. The air was turned on when the colonoscope reached the cecum.
  Interventions: Procedure: water exchange
- cap-assisted water exchange (Experimental): Cap was mounted to the tip of the colonoscope when water exchange was performed.
  Interventions: Device: cap-assisted water exchange; Procedure: water exchange

INTERVENTIONS:
Device: cap-assisted water exchange — a transparent cap was mounted to the tip of colonoscopy when water exchange was performed.
  Arms: cap-assisted water exchange
Procedure: water exchange — water was infused and suctioned at the same time during insertion of colonoscope

SUMMARY:
This prospective, randomize, controlled trial will compared cap-assisted water exchange with water exchange in patients undergoing sedated colonoscopy. Investigators test the hypothesis that that cap-assisted water exchange is more efficient and causes a shorter insertion time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing fully sedated colonoscopy performed by the investigators

Exclusion Criteria:

* obstructive lesions of the colon
* massive ascites
* history of partial colectomy
* provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
cecal intubation time | when the colonoscope reaches the cecum, an average of 14 minutes

SECONDARY OUTCOMES:
Dose of propofol | The end of colonoscopy, an average of 14 minutes
adenoma detection rate | One week after colonoscopy
  when histology analysis of the removed polyps are available

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, MD, Principal Investigator — Dalin Tzu Chi Hospital. Tzu Chi medication Foundation
Locations (1):
- Dalin Tzu Chi General Hospital, Chiayi City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung FW, Amato A, Ell C, Friedland S, Harker JO, Hsieh YH, Leung JW, Mann SK, Paggi S, Pohl J, Radaelli F, Ramirez FC, Siao-Salera R, Terruzzi V. Water-aided colonoscopy: a systematic review. Gastrointest Endosc. 2012 Sep;76(3):657-66. doi: 10.1016/j.gie.2012.04.467. PMID 22898423
- [Background] Rastogi A, Bansal A, Rao DS, Gupta N, Wani SB, Shipe T, Gaddam S, Singh V, Sharma P. Higher adenoma detection rates with cap-assisted colonoscopy: a randomised controlled trial. Gut. 2012 Mar;61(3):402-8. doi: 10.1136/gutjnl-2011-300187. Epub 2011 Oct 13. PMID 21997547
- [Background] Kondo S, Yamaji Y, Watabe H, Yamada A, Sugimoto T, Ohta M, Ogura K, Okamoto M, Yoshida H, Kawabe T, Omata M. A randomized controlled trial evaluating the usefulness of a transparent hood attached to the tip of the colonoscope. Am J Gastroenterol. 2007 Jan;102(1):75-81. doi: 10.1111/j.1572-0241.2006.00897.x. Epub 2006 Nov 13. PMID 17100978
- [Background] Lee YT, Lai LH, Hui AJ, Wong VW, Ching JY, Wong GL, Wu JC, Chan HL, Leung WK, Lau JY, Sung JJ, Chan FK. Efficacy of cap-assisted colonoscopy in comparison with regular colonoscopy: a randomized controlled trial. Am J Gastroenterol. 2009 Jan;104(1):41-6. doi: 10.1038/ajg.2008.56. PMID 19098847